CLINICAL TRIAL: NCT01967836
Title: Glad Press 'n Seal® as a Temporary Moisture Barrier to Central Lines in Ambulatory Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen T Greene (Other)
Responsible Party: Sponsor-Investigator, Maureen T Greene, Maureen T. Greene, PhD, RN, Wheaton Franciscan Healthcare
Organization: Wheaton Franciscan Healthcare (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-059
Record Dates: First submitted 2013-10-07; First posted 2013-10-23 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Cancer-related Problem/Condition; Ambulatory Care
Keywords: Invasive Line; IV Dressing protection; Hygiene; Oncology; Ambulatory Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glad Press 'n Seal (Other): Cohort Subjects will use Glad Press 'n Seal product as a moisture barrier to an IV line
  Interventions: Device: Glad Press 'n Seal

INTERVENTIONS:
Device: Glad Press 'n Seal — Application of Glad Press n' Seal product as an IV site dressing protection during subject showering

SUMMARY:
The purpose of this study is to see if Glad Press 'n Seal works as a moisture barrier for central line that is left in place during ambulatory oncology clinical care.

DETAILED DESCRIPTION:
Enrolled subjects will be instructed on the application of the Glad Press 'n Seal product to their IV dressing for use during a shower activity. Practice with application and removal of the product will be supervised by the PI or RA. Questions will be answered and a commercially purchased box of the investigational product will be given to the subject for home use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring mediport or peripherally inserted central venous catheter line access for 3-5 days
* Able to read and write English
* Use showering as a means of home hygiene

Exclusion Criteria:

* Subjects with eczema/psoriasis at the line insertion area
* Subjects with active line/site irritation/infection
* Subjects on chemotherapy protocols including anti-epidermal growth factor receptor drugs (cetuximab, panitumumab) or ipilimumab as there is a high incidence of skin rash as a side effect of these medications
* Patients who do not intend to shower as a means of home hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen T Greene, PhD, RN, Principal Investigator — Wheaton Franciscan Healthcare
Locations (4):
- United States (4):
  - Rieman Cancer Center, Milwaukee, Wisconsin
  - Wheaton Franciscan Healthcare-St Joseph campus, Milwaukee, Wisconsin
  - WFH-St. Francis, Milwaukee, Wisconsin
  - Wheaton Franciscan - Wauwatosa Campus, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Glad Press 'n Seal: Subjects will use Glad Press 'n Seal product as a moisture barrier to an IV line
  Glad Press 'n Seal: Application of Glad Press n' Seal product as an IV site dressing protection during subject showering as a means of bathing
Period: Overall Study
Arm/Group | Glad Press 'n Seal
Started | 20
Completed | 11
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Subjects who present to ambulatory oncology or outpatient clinic sites with the presence of a centrally placed IV catheter for infusion therapy who meet were approached for consent
  19 Oncology subjects who met criteria were approached with 9 declines to participate 1 ambulatory care subject was approached and accepted participation
Groups:
- Glad Press 'n Seal: Subjects will use Glad Press 'n Seal product as a moisture barrier to an IV line
  Glad Press 'n Seal: Application of Glad Press n' Seal product as an IV site dressing protection during subject showering
Arm/Group | Glad Press 'n Seal
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
subjects with central IV catheter in place [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Subject Questionnaire Post Shower Evaluation
Description: Percentage of responses to evaluation questions (Percentage reported are "yes" responses) for the following questions. 40 surveys were returned from 11 patient subjects.
  1. Did you need assistance to place the Glad Press 'n Seal to your IV area?
  2. Was the area covered by the Glad Press 'n Seal dry after taking it off?
  3. Was the dressing covering your IV undamaged after taking off the Glad Press 'n Seal?
  4. Did you feel the IV Line was accidentally pulled at all with the use of the Glad Press 'n Seal?
  Likert Scale response to the following question On a scale of 0 (would not use) to 10 (would continue to use) how satisfied were you in using Glad Press n Seal?
Time Frame: complete one evaluation after each shower when using product
Population: 10 oncology and 1 ambulatory subjects returned 39 evaluation forms for primary analysis
Measure: Number; unit: percentage of yes responses
Groups:
- Glad Press 'n Seal: Subjects will use Glad Press 'n Seal product as a moisture barrier to an IV line
  Glad Press 'n Seal: Application of Glad Press n' Seal product as an IV site dressing protection during subject showering.
  Subject specific characteristics 19 subjects in oncology clinic sites were approached to participate; 9 refused participation
  1 subject in ambulatory clinic was approached and was consented
Arm/Group | Glad Press 'n Seal
Number analyzed (Participants) | 11
percentage of yes responses
  Question 1 | 80
  Question 2 | 88
  Question 3 | 76
  Question 4 | 0

2. Primary Outcome: Patient Satisfaction Mean on a 0-10 Likert Scale on the Use of Glad Press 'n Seal During Showering. 40 Subjects Reports.
Description: 0 Not at all satisfied 10 Very satisfied
Time Frame: Reported afer each subject showering survey completion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glad Press 'n Seal
Number analyzed (Participants) | 11
units on a scale | 7.65 (2.91)

3. Secondary Outcome: Clinic Nurse Observation of Subjects, Who Used Intervention Device, at the Next Clinic Visit
Description: The secondary outcomes of the study are clinic nurse observed problems. Percentage of "yes" responses of nurse observations of site at clinic visit
  1. Line dressing intact (Yes) is in place (reporting on 20 lines on 28 RN observations)
  2. Absence (No) of local skin irritation,
  3. Dislodgement of the IV line/needle (No) with the IV site upon subject return to the clinic and verification by the subject .
Time Frame: Inspection of central line site and dressing upon return to schduled clinic visit up to 30 days
Population: Nurse questionnaire evaluation forms were completed relative to subjects questionnaires being returned at next clinic visit
Measure: Number; unit: percentage of observation
Units Other Than Participants: Nurse Observation of IV Site
Groups:
- Glad Press 'n Seal: Subjects will use Glad Press 'n Seal product as a moisture barrier to an IV line
  Glad Press 'n Seal: Application of Glad Press n' Seal product as an IV site dressing protection during subject showering.
  Subject specific characteristics 19 subjects in oncology clinic sites were approached to participate; 9 refused participation
  1 subject in ambulatory clinic was approached and was consented
  Nurses inspection of central line site on study participants at next clinic visit with return of subject patient questionnaire evaluation of use of product device with showing 27 nurse evaluations were completed for analysis
Arm/Group | Glad Press 'n Seal
Number analyzed (Participants) | 11
Number analyzed (Nurse Observation of IV Site) | 28
percentage of observation
  Nurse Question 1 | 91
  Nurse Question 2 | 93
  Nurse Question 3 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Description: Only pre-specified to monitor for device related adverse events
Arm/Group | Glad Press 'n Seal
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes